CLINICAL TRIAL: NCT07039162
Title: Phase II Study of Tislelizumab Combined With Induction Chemoradiotherapy and Subsequent Conversion Surgery for Locally Advanced Unresectable ESCC
Brief Title: Study of Tislelizumab Combined With Chemoradiotherapy and Surgery for Unresectable Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ming-Yu Lien (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor-Investigator, Ming-Yu Lien, Department of Hematology and Oncology, China Medical University Hospital, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH-BGB-A317-CS01
Record Dates: First submitted 2025-06-11; First posted 2025-06-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC); Locally Advanced Unresectable Esophageal Cancer
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; Paclitaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Single-arm study: Participants will receive Tislelizumab in combination with chemoradiotherapy (Paclitaxel + Cisplatin) and conversion surgery if the tumor becomes resectable. The treatment sequence involves induction chemoradiotherapy, followed by consolidation chemotherapy and surgery if applicable.
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Tislelizumab — 1. ICRT phase -Tislelizumab and CRT regimen Tislelizumab 200 mg IV, C1D1 and C4D1
  2. Consolidation phase: Tislelizumab-Paclitaxel-Cisplatin regimen Tislelizumab 200 mg IV, D1, every 3 weeks (*The regimen is repeated until unacceptable toxicity or disease progression, up to maximum of 2 cycles. )
  3. Adjuvant phase-Tislelizumab Tislelizumab 200 mg IV, D1, every 3 weeks (*The regimen is repeated until unacceptable toxicity or disease progression, up to maximum of one year or 17 cycles.)
Drug: Paclitaxel — 1. ICRT phase -Tislelizumab and CRT regimen Paclitaxel 50 mg/m2 IV, D1, weekly (* 4-6 cycles judged by investigators.)
  2. Consolidation phase: Tislelizumab-Paclitaxel-Cisplatin regimen Paclitaxel 135 mg/m2 IV, D1, every 3 weeks (*The regimen is repeated until unacceptable toxicity or disease progression, up to maximum of 2 cycles.)
Drug: Cisplatin — 1. ICRT phase -Tislelizumab and CRT regimen Cisplatin 25 mg/m2 IV, D1, weekly ( 4-6 cycles judged by investigators.)
  2. Consolidation phase: Tislelizumab-Paclitaxel-Cisplatin regimen Cisplatin 75 mg/m2 IV, D1, every 3 weeks (*The regimen is repeated until unacceptable toxicity or disease progression, up to maximum of 2 cycles. )
Radiation: Radiation Therapy — 1. ICRT phase -Tislelizumab and CRT regimen Radiotherapy treatment: IMRT 41-50.4Gy, a dose of 1.8 to 2Gy per day, 5 days per week for 5 weeks during the RT phase.

SUMMARY:
This is a Phase II, open-label, single-arm, multicenter study evaluating the safety and efficacy of combining Tislelizumab with induction chemoradiotherapy (CRT), followed by conversion surgery, in patients with locally advanced, unresectable esophageal squamous cell carcinoma (ESCC).

Patients will receive induction CRT with weekly paclitaxel and cisplatin along with Tislelizumab, followed by two cycles of consolidation Tislelizumab-chemotherapy. If the tumor becomes resectable, patients will undergo surgery.

The primary goal is to assess the 2-year overall survival (OS) rate. Secondary outcomes include pathological complete response (pCR), conversion rate, R0 resection rate, disease-free survival (DFS), recurrence-free survival (RFS), and treatment-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had histologically confirmed, squamous-cell carcinoma of the esophagus
2. Clinical T4 cancer, at least one unresectable metastatic regional lymph node due to invasion into an adjacent organ, or computed tomographic (CT) evidence of M1Lym, such as fixed supraclavicular nodes. Regional lymph nodes are defined on the basis of criteria specified by the eighth edition of the Union for International Cancer Control TNM staging system (Sobin and Wittekind, 2016).
3. An age of at least 20 years
4. An Eastern Cooperative Oncology Group performance-status score 0 or 1
5. Adequate major organ functions

   * WBC ≥3,500/mm3
   * Hemoglobin ≥ 9.0 g/dL
   * Platelet ≥ 80,000/mm3
   * Total bilirubin ≤ 2-fold the upper limit of normal (ULN)
   * ALT and AST ≤ 5-fold the ULN AND ≤200 U/L
   * PT, aPTT and INR ≤1.5-fold the ULN
   * Albumin ≥2.5 g/dL
   * Creatinine clearance ≥50 ml/min (based upon 24 hours urine collection or calculated by Cockroft-Gault formula)

     * Male: ((140 - age) × weight [kg])/(72 × serum creatinine [mg/dL])
     * Female: 0.85 x estimate for male
6. Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons) must agree to use contraception from the time of informed consent until 5 months or more after the last dose of investigational products. (Women of childbearing potential are defined as all women after the onset of menstruation who are not postmenopausal and have not been surgically sterilized (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy). Postmenopause is defined as amenorrhea for ≥12 consecutive months without specific reasons.)
7. Men must agree to use contraception from the start of study treatment until 3 months or more after the last dose of the investigational product.
8. Patients must be willing to undergo definitive resection with lymph node dissection
9. Participants must have signed written informed consent form in accordance with regulatory and institutional guidelines.

Exclusion Criteria:

1. Patient has received systemic therapy for advanced ESCC.
2. Patients had distant metastasis, including liver, lung, bone and brain metastases.
3. Patients had esophageal perforation or esophageal fistula
4. Patients had tumor bleeding
5. Patients had active infection(e.g. tuberculosis).
6. History or known human immunodeficiency virus.
7. Subjects with active, known, or suspected autoimmune disease. Subjects with Type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll.
8. Systemic immunosuppression therapy or chronic systemic steroid therapy (more than 10mg daily of prednisolone)
9. Known hepatitis B (HBsAg reactive) or C virus infection (positive anti HCV)

   * Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA < 500 IU/mL or < 2500 copies/mL) can be enrolled. Patients with detectable HBsAg or detectable HBV DNA should be managed per treatment guidelines. Patients receiving antivirals at screening should have been treated for > 2 weeks before randomization/enrollment.
   * Patients with a positive HCV antibody test followed by a negative HCV RNA test at screening are eligible.
10. Previous therapy targeting T-cell costimulating or immune-checkpoint pathways
11. Prior or concurrent malignancies within the last 3 years, with the exception of carcinoma in situ of the cervix, or basal type skin cancer
12. Any major surgery within 4 weeks before study enrollment.
13. Pregnant women or nursing mothers, or positive pregnancy tests
14. Patients had allogeneic stem cell transplantation or organ transplantation.
15. Has uncontrolled, significant cardiovascular disease or cerebrovascular disease, including NYHA Class III or IV congestive heart failure, unstable angina, myocardial infarction, uncontrolled symptomatic arrhythmia, and/or other serious cardiovascular and cerebrovascular diseases within the 6 months preceding study intervention.
16. Patients with interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases including pulmonary fibrosis, or acute lung diseases
17. Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
18. Other patients judged by the investigators be inappropriate as subjects of this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year OS rate | From the date of first treatment (induction chemoradiotherapy) to 2 years after treatment initiation.
  Estimated 2-year OS rate is defined as number of participants alive divided by the number of participants.

SECONDARY OUTCOMES:
Pathological complete response (pCR) rate | At time of surgery (8 to 12 weeks after completion of induction or consolidation treatment)
  Pathological complete response (pCR) rate is defined as number of participants with no evidence of residual tumor cells in the primary site and resected lymph nodes of the operative specimens divided by the number of participants received esophagectomy.
Conversion rate | Assessed within 12 weeks after completion of induction or consolidation treatment.
  Conversion rate is defined asnumber of participants received esophagectomy divided by the number of participants.
R0 resection rate | Assessed at time of surgery (8 to 12 weeks after completion of induction or consolidation treatment)
  R0 resection rate is defined as the proportion of participants with negative resection margins (greater than 1 mm) among those who underwent esophagectomy following induction chemoradiotherapy and/or consolidation treatment with tislelizumab.
Disease-free survival (DFS) | From enrollment until disease recurrence or death, whichever occurs first, assessed up to 2 years.
  Disease-free survival (DFS) is defined as the time from enrollment until evidence of disease recurrence or death.
Event-free survival (EFS) | From date of enrollment to first documented event or death, assessed up to 2 years.
  Event-free survival (EFS) is defined as the time from enrollment to an event which may include radiographic progression, clinical progression, 2nd aerodigestive tract squamous cell carcinoma, and death.
Distant metastasis-free survival (DMFS) | From date of enrollment to first documented distant metastasis or death, assessed up to 2 years
  Distant metastasis-free survival (DMFS) is defined as the time from enrollment until evidence of distant metastasis recurrence or death.
Overall survival (OS) | From date of enrollment to death, assessed up to 2 years
  Overall survival (OS) is defined as the time from enrollment to death
Recurrence-free survival (RFS) | From date of initial treatment to first documented recurrence or death, assessed up to 2 years
  Recurrence-free survival (RFS) is Measure the length of time that patients remain free of disease recurrence or progression following initial treatment.
Adverse events | From the date of informed consent until the completion of study treatment and follow-up period, up to 2 years.
  Adverse events related to protocol immunotherapy, chemotherapy, radiotherapy and conversion surgery .

CONTACTS AND LOCATIONS:
Locations (7):
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District